CLINICAL TRIAL: NCT05034523
Title: Voxel Based Morphometry In Patients With Psychotic Versus Non Psychotic Depression
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Doaa Noor Eldin Abdelazeem Mohammed, Assistant lecturer, Assiut University
Other Study IDs: Voxel based MRI in depression
Record Dates: First submitted 2021-08-24; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Psychotic Depression; Non Psychotic Depression
Keywords: Depression; Psychotic depression; Voxel based morphometry
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: MRI Voxel based morphometry — Voxel based morphometry through analysis of 3D T1 weighted sequence to assess total intracranial volume. All participants were scanned on the 1.5Tesla MR scanner (Achieva, Philips Medical Systems, Best, NL) with a 16-channel head coil at the diagnostic radiology department.

SUMMARY:
1. To examine structural brain changes in patients with depression measured using voxel based morphometry(VBM) in comparison with healthy subjects.
2. Relation between grey mater volume (GMV) and other structural changes, and the severity of clinical symptoms.
3. To study if there is structural brain difference between psychotic and non-psychotic depression

DETAILED DESCRIPTION:
Depression is a major psychiatric disorder and a leading cause of disability worldwide. The clinical representation encompasses affective, cognitive and somatic complains such as low mood, anxiety, lack of pleasure and interest, disturbances of sleep and appetite, decreased self-esteem, thoughts of guilt, hopelessness, and even suicide.

Major depressive disorder (MDD) with psychotic features (psychotic depression) is a severe disorder with a lifetime prevalence of 0.35-1% .

Over the last decades, increasing evidence from post-mortem studies and in vivo studies emerged that mood disorder can induce structural and morphometric changes of the brain The development of magnetic resonance imaging (MRI) has allowed for more advanced structural imaging

Several structural magnetic resonance imaging (s MRI) studies have identified key brain areas involved in MDD. In particular, voxel-based morphometry (VBM), it is helpful in quantitatively identifying unexpected anatomic changes studies have found that MDD is associated with widespread local brain abnormalities, mainly affecting the frontal gyrus, insula, temporal lobes and anterior cingulate gyrus . Structural white matter alterations have also been reported within the inferior parietal lobule and frontal gyrus .

Many studies are positive about grey matter (GM) volume reductions in various cortical regions in depressed patients compared to healthy controls . The most consistent findings appear to be related to GM loss in medial frontal cortex (MFC), anterior cingulate cortex (ACC) and orbitofrontal cortex (OFC) with less evidence about subcortical structures such as the amygdala and the hippocampus .

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60 years old.
2. Based on DSM5 Criteria: MDD with or without psychotic features.

Exclusion Criteria:

1 • Patients under 18 years old or above 60

2• Pregnant or lactating women.

3• Other current or past major psychiatric disorders

4• History or concurrent neurological disease(seizures) or prior head trauma with evidence of consequent cognitive impairment.

5• First degree family history of schizophrenia if the participant is less than 33 years old (mean age of onset of schizophrenia plus two standard deviations) to exclude possible prodromal phase of schizophrenia.

6• Unstable medical condition (i.e., any active illness that may affect the brain as blood dyscrasis, lymphomas, endocrinopathies, renal failure, chronic obstructive lung disease, systemic autoimmune disorders or Malignancy).

7• Patients being treated with steroids or hormonal therapy .

8• Current substances or alcohol use disorders (past diagnosis allowed if in remission for more than 6 months

9• Contraindications for MRI as:

* Metal implants or paramagnetic objects contained within the body (including heart pacemaker or surgical prosthesis)
* Claustrophobia significant enough to interfere with MRI

  10• Refusal of informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study included two groups:
  Group (A): patients' group diagnosed with major depressive disorder (MDD) which include (44) patients aged 18-60 years' old who attended psychiatric outpatient's clinic and who is admitted in psychiatric unit of Assiut university hospitals. This group is further subdivided according to DSM 5 Criteria into 2 subgroups: Major depression with psychotic disorder and Major depression without psychotic disorder.
  Group (B): control group which consists of (22) healthy cross matching individuals.
Sampling Method: Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Study the structural brain changes in different areas in patients with psychotic depression and non-psychotic depression. | one year
  Investigators will use MRI the voxel based morphometry to measure the volume of different areas in grey and white matter in depressed patients and compare them to structure of brain in healthy group.
Examine different variables related to major depressive disorder and their specific relation to structural changes in different areas in brain | one year
  Investigators will measure the changes occur in volume of different areas in brain with different types of depression.
  Investigators will measure the changes in volume of different areas in brain which occur by the effect of psychotic features.
  Investigators will measure the effect of suicide on changes of volume of different areas of brain.

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Elserogy, MD, Study Chair — Assiut University

REFERENCES:
- [Background] Sacher J, Neumann J, Funfstuck T, Soliman A, Villringer A, Schroeter ML. Mapping the depressed brain: a meta-analysis of structural and functional alterations in major depressive disorder. J Affect Disord. 2012 Oct;140(2):142-8. doi: 10.1016/j.jad.2011.08.001. Epub 2011 Sep 3. PMID 21890211
- [Background] Jaaskelainen E, Juola T, Korpela H, Lehtiniemi H, Nietola M, Korkeila J, Miettunen J. Epidemiology of psychotic depression - systematic review and meta-analysis. Psychol Med. 2018 Apr;48(6):905-918. doi: 10.1017/S0033291717002501. Epub 2017 Sep 12. PMID 28893329
- [Background] Lui S, Zhou XJ, Sweeney JA, Gong Q. Psychoradiology: The Frontier of Neuroimaging in Psychiatry. Radiology. 2016 Nov;281(2):357-372. doi: 10.1148/radiol.2016152149. PMID 27755933
- [Background] O'Connor S, Agius M. A systematic review of structural and functional MRI differences between psychotic and nonpsychotic depression. Psychiatr Danub. 2015 Sep;27 Suppl 1:S235-9. PMID 26417770
- [Background] Schmaal L, Veltman DJ, van Erp TG, Samann PG, Frodl T, Jahanshad N, Loehrer E, Tiemeier H, Hofman A, Niessen WJ, Vernooij MW, Ikram MA, Wittfeld K, Grabe HJ, Block A, Hegenscheid K, Volzke H, Hoehn D, Czisch M, Lagopoulos J, Hatton SN, Hickie IB, Goya-Maldonado R, Kramer B, Gruber O, Couvy-Duchesne B, Renteria ME, Strike LT, Mills NT, de Zubicaray GI, McMahon KL, Medland SE, Martin NG, Gillespie NA, Wright MJ, Hall GB, MacQueen GM, Frey EM, Carballedo A, van Velzen LS, van Tol MJ, van der Wee NJ, Veer IM, Walter H, Schnell K, Schramm E, Normann C, Schoepf D, Konrad C, Zurowski B, Nickson T, McIntosh AM, Papmeyer M, Whalley HC, Sussmann JE, Godlewska BR, Cowen PJ, Fischer FH, Rose M, Penninx BW, Thompson PM, Hibar DP. Subcortical brain alterations in major depressive disorder: findings from the ENIGMA Major Depressive Disorder working group. Mol Psychiatry. 2016 Jun;21(6):806-12. doi: 10.1038/mp.2015.69. Epub 2015 Jun 30. PMID 26122586
- [Background] Yuan Y, Zhang Z, Bai F, Yu H, You J, Shi Y, Qian Y, Liu W, Jiang T. Larger regional white matter volume is associated with executive function deficit in remitted geriatric depression: an optimized voxel-based morphometry study. J Affect Disord. 2009 May;115(1-2):225-9. doi: 10.1016/j.jad.2008.09.018. Epub 2008 Oct 21. PMID 18945494
- [Background] Lai CH. Gray matter volume in major depressive disorder: a meta-analysis of voxel-based morphometry studies. Psychiatry Res. 2013 Jan 30;211(1):37-46. doi: 10.1016/j.pscychresns.2012.06.006. Epub 2012 Nov 10. PMID 23146253
- [Background] Arnone D, Job D, Selvaraj S, Abe O, Amico F, Cheng Y, Colloby SJ, O'Brien JT, Frodl T, Gotlib IH, Ham BJ, Kim MJ, Koolschijn PC, Perico CA, Salvadore G, Thomas AJ, Van Tol MJ, van der Wee NJ, Veltman DJ, Wagner G, McIntosh AM. Computational meta-analysis of statistical parametric maps in major depression. Hum Brain Mapp. 2016 Apr;37(4):1393-404. doi: 10.1002/hbm.23108. Epub 2016 Feb 8. PMID 26854015